CLINICAL TRIAL: NCT01416090
Title: Syndactyly Repair: Comparison of Skin Graft and No Skin Graft Techniques
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, M.D., University of Utah
Other Study IDs: 12534
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Congenital Hand Deformities
Keywords: syndactyly
MeSH Terms: conditions — Hand Deformities, Congenital; Syndactyly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Syndactyly is a relatively common congenital abnormality of the hand occurring approximately 1 out of 2500 live births (1). It can be simple, meaning only skin and soft tissues are shared, or complex, meaning the bone or nail parts are shared. In any case, it is a fact that there is not enough skin surrounding the two finger segment to be utilized to cover two separate fingers. This can also be proven by simple geometry. Therefore, it has always been taught to residents and explained to numerous patients' families that addition of skin graft is required for a proper syndactyly release. Without it, skin flaps would be too tight, causing some necrosis and significant scarring along the finger and particularly in the web space, causing an unsatisfactory functional and cosmetic result requiring revision.

DETAILED DESCRIPTION:
Syndactyly is a relatively common congenital abnormality of the hand occurring approximately 1 out of 2500 live births (1). It can be simple, meaning only skin and soft tissues are shared, or complex, meaning the bone or nail parts are shared. In any case, it is a fact that there is not enough skin surrounding the two finger segment to be utilized to cover two separate fingers. This can also be proven by simple geometry. Therefore, it has always been taught to residents and explained to numerous patients' families that addition of skin graft is required for a proper syndactyly release. Without it, skin flaps would be too tight, causing some necrosis and significant scarring along the finger and particularly in the web space, causing an unsatisfactory functional and cosmetic result requiring revision.

Full thickness skin grafts (FTSG) are usually utilized for this procedure and come at some cost. An additional incision, and therefore scar, is made in the groin or on the arm or hand itself. The skin graft itself usually has a slightly different color and further hyperpigments (2, 3, 4, 5) when placed on the hand and can have hair growth that would not normally be present between fingers. These create cosmetic issues as the patient gets older. In addition, skin graft is quite cumbersome to utilize in these tight areas and small fingers of small children. It definitely adds to the time under anesthesia because no method other than sewing with small sutures has been shown to be efficacious. Whereas the release of a simple syndactyly may take 30-60 minutes, the suturing of skin graft and the skin flaps usually takes one and half times that long in addition. Further, skin grafts require immobilization and special bandaging techniques to avoid graft loss. One final disadvantage of full thickness skin grafts is that they have been implicated in the occurrence of web creep, which is a post-operative scarring between fingers that decreases the amount of web space originally obtained (4,6). These will often require further surgical procedures (Percival & Sykes).

Over the last 20 years, there has been resurgence in attempts to treat syndactyly without skin grafts (8, 9, 10, 11, 12, 3, 6). All techniques include a significant defatting of the subcutaneous tissues all the way back to the web space in an effect to decrease circumference of the digits. Different dorsal metacarpal flaps have been described as well, including local island pedicle flaps that can be used for the web commissure (3, 9, 10, 11). In addition, it has been shown that leaving flaps slightly open, up to 2mm, for secondary intention healing creates good scars in children and no increased sign of web creep or flexion contracture (5). Combining all three of these techniques leads to the technical ability of syndactyly release without the need for skin grafts. Proven benefits have been the lack of the donor scar, lack of pigmented or hairy graft sites, and decreased operative time. However, the incidences of web creep, flexion or lateral contractures, reoperation rate and the final cosmetic result have not been proven to be better or worse, as no one has compared similar patients. All studies to date have been instead a review of results using their particular technique that does not require skin graft. If any comparisons have been made, it has been using historical data already published.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6 months to 6 years with simple syndactyly 2nd and/or 3rd web space without other major congenital hand abnormally syndrome that would affect growth, function, and appearance of hand.

Exclusion Criteria:

* patients with complex syndactyly, syndactyly of teh first web, patients with brachysyndactyly and diagnosis of Apert's, poland's and other syndromes that often include incomplete digital components and subsequent function.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Syndactyly is a relatively common congenital abnormality of the hand occurring approximately 1 out of 2500 live births. We will utilize children under the age of 6 years and over the age of 6 months. Most will likely be less than 2.5 years of age. This surgery is usually performed when the patient is still a child.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2004-07; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
compare this newer technique to the gold standard full thickness skin graft technique | 5 years
  Patients will all be treated with the same post-operative dressing and the same post-operative protocol. They will be followed in the same manner, approximately one month from surgery when the dressings will be removed, three months from surgery and then yearly. Final assessment, including the objective testing of their fingers, will be performed by an independent therapist experienced in congenital pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas T Hutchinson, M.D., Principal Investigator — University of Utah Orthopedic Center
Locations (1):
- University of Utah Orthopedic Center, Salt Lake City, Utah, United States